CLINICAL TRIAL: NCT00540059
Title: Quality Assurance Project in Patients With Advanced Prostate Carcinoma - Evaluation of Tolerability, Quality of Life and Usage of Zoladex 10,8 SafeSystem
Brief Title: Evaluation of QoL, Tolerability and Use of Zoladex 10,8 SafeSystem for Advanced PCa - German IPEP Trial
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: Zx-002
Record Dates: First submitted 2007-10-03; First posted 2007-10-05 (Estimated); Last update posted 2007-10-05 (Estimated); Status verified 2007-08

CONDITIONS: Prostate Carcinoma
Keywords: Prostate carcinoma; LHRH; Zoladex
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Purpose of this study is the evaluation of QoL, tolerability and use of Zoladex 10,8 SafeSystem for advanced PCa under naturalistic conditions

ELIGIBILITY:
Inclusion Criteria:

* Patients with PCa, who will be treated with Zoladex 10,8 SafeSystem based on the current SPC

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1950 (Actual)
Dates: Start 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: H Brasch, Study Director — AstraZeneca